CLINICAL TRIAL: NCT01458574
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Of Oral Cp-690,550 As A Maintenance Therapy In Subjects With Ulcerative Colitis
Brief Title: A Study Of Oral CP-690,550 As A Maintenance Therapy For Ulcerative Colitis
Acronym: OCTAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3921096; 2011-004580-79 (EudraCT Number); OCTAVESUSTAIN (Other: Alias Study Number)
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Ulcerative Colitis
Keywords: Janus kinase inhibitor; JAK 3 inhibitor; inflammatory bowel disease; ulcerative colitis; OCTAVE; CP-690; 550; tofacitinib; Xeljanz
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo
- CP-690,550 5 mg Arm (Experimental)
  Interventions: Drug: CP690,550
- CP-690,550 10 mg Arm (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: Placebo — Placebo 10 mg orally (PO) twice a day (BID)
  Arms: Placebo Comparator
Drug: CP690,550 — CP-690,550 5 mg orally (PO) twice a day (BID)
  Arms: CP-690,550 5 mg Arm
Drug: CP-690,550 — CP-690,550 10 mg orally (PO) twice a day (BID)
  Arms: CP-690,550 10 mg Arm

SUMMARY:
The study proposes to assess whether compared to placebo, CP-690,550 is effective, safe, and tolerable maintenance therapy in subjects with Ulcerative Colitis (UC). The study proposes to assess whether compared to placebo, CP-690,550 maintenance therapy more effectively achieves mucosal healing and improves quality of life in subjects with UC.The study proposes to assess CP-690,550 pharmacokinetic exposure during maintenance therapy in subjects over the age of 18 years with UC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who met study entry criteria and completed 8-week induction treatment from Study A3921094 or A3921095
* Subjects who achieved clinical response in Study A3921094 or A3921095
* Women of childbearing potential must test negative for pregnancy prior to study enrollment
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Evidence of a personally signed and dated informed consent document(s) indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Subjects who had major protocol violation (as determined by the Sponsor) in Study A3921094 or A3921095
* Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, or clinical findings suggestive of Crohn's disease
* Subjects who have had surgery for UC or in the opinion of the investigator, are likely to require surgery for UC during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2012-07-20 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (274):
- United States (94):
  - Internal Medicine Center, LLC, Mobile, Alabama
  - Springhill Memorial Hospital (Endoscopy Only), Mobile, Alabama
  - UCSD Health System - Investigational Drug Pharmacy - Moores Cancer Center, La Jolla, California
  - UCSD Medical Center, La Jolla, California
  - Alliance Clinical Research, Oceanside, California
  - Desert Advanced Imaging, Palm Springs, California
  - Erik Palmer, DO, Palm Springs, California
  - Homan A Zadeh, MD, MPH, Palm Springs, California
  - Hope Square Surgical Center, Rancho Mirage, California
  - Sharp Rees-Stealy Medical Group, Inc., San Diego, California
  - Clinical Applications Laboratories, Inc, San Diego, California
  - San Diego Endoscopy Center, San Diego, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - UCSF Endoscopy Unit at Mount Zion, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Bristol Hospital, Bristol, Connecticut
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Endoscopy Center of Connecticut, LLC, Guilford, Connecticut
  - Endoscopy Center of Connecticut, LLC, Hamden, Connecticut
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Central Connecticut Endoscopy Center, Plainville, Connecticut
  - Citrus Surgery & Endoscopy Center (colonoscopy), Crystal River, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Suncoast Endoscopy Center (colonoscopy), Inverness, Florida
  - North Florida Gastroenterology Research, LLC, Orange Park, Florida
  - Citrus Ambulatory Surgery Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Advanced Gastroenterology Center, Port Orange, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Endoscopy Center, Port Orange, Florida
  - Port Orange Urgent Care, Port Orange, Florida
  - Florida Medical Clinic, P.A., Zephyhills, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Georgia Endoscopy Center, Alpharetta, Georgia
  - GI Consultants, Atlanta, Georgia
  - Emory Healthcare Heart Center, Johns Creek, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Johns Creek Diagnostic Center, Suwanee, Georgia
  - Cotton-O'Neal Clinical Research Center Digestive Health, Topeka, Kansas
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Gastrointestinal Diagnostic Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Howard County GIDC, Columbia, Maryland
  - Saint Joseph Mercy Hospital - Inpatient Pharmacy, Ann Arbor, Michigan
  - East Ann Arbor Health and Geriatrics Center - UMHS, Ann Arbor, Michigan
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Michigan Clinical Research Unit - UMHS, Ann Arbor, Michigan
  - Medical Science Research Building 1 - UMHS, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Surgical Centers of Michigan, Troy, Michigan
  - Utica Surgery Center (Endoscopy Only), Utica, Michigan
  - Michigan Heart SJMH, Ypsilanti, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Saint Joseph Mercy Hospital Outpatient Laboratory, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - AGA Clinical Research Associates, LLC, Egg Harbour Township, New Jersey
  - South Jersey Gastroenterology, Marlton, New Jersey
  - The Endo Center at Voorhees, Vorhees, New Jersey
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - NYU Langone Nassau Gastroenterology Associates, Great Neck, New York
  - The Private Practice of Simon Lichtiger, MD, New York, New York
  - IBD Center - The Mount Sinai Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - CUMC Research Pharmacy, New York, New York
  - Kornbluth, Legnani, George MD, PC, New York, New York
  - University of Rochester, Rochester, New York
  - Carolina Research, Carolina Digestive Diseases, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Mentor Medical Campus, Mentor, Ohio
  - The Endoscopy Center of Lake County, Mentor, Ohio
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Professional Quality Research, Inc.- Austin Gastroenterology PA, Austin, Texas
  - Austin Endoscopy Center II, Austin, Texas
  - Austin Gastroenterology PA, Austin, Texas
  - Houston Hospital for Specialized Surgery (Endoscopy only), Houston, Texas
  - Baylor College of Medicine (Baylor Medical Center), Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center (Drug Storage), Houston, Texas
  - McGovern Medical School -The University of Texas Health Science Center at Houston, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Alpine Medical Group, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Wasatch Endoscopy Center, Salt Lake City, Utah
  - VCU Health System Digestive Health Center, Richmond, Virginia
  - VCU Health System Endoscopy Suite, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - The Center for Digestive Health, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Eastern Health-Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
- AKH Wien, Universitaetsklinik fuer Innere Medizin III, Vienna, Vienna, Austria
- Belgium (4):
  - GZA St. Vincentius, Antwerp
  - AZ Groeninge, Kortrijk
  - UZ Leuven (University Hospital Leuven), Campus Gasthuisberg, Leuven
  - H-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Hospital de Clinicas de Porto Alegre - HCPA, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (7):
  - University of Alberta Hospital - Walter C. Mackenzie Health Sciences Centre, Edmonton, Alberta
  - University of Alberta - Zeidler Ledcor Centre, Edmonton, Alberta
  - McMaster University Medical Center, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
- Instituto de Coloproctología ICO S.A.S., Medellín, Antioquia, Colombia
- University Hospital Center Zagreb, Zagreb, Croatia
- Czechia (3):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Nemocnice Strakonice, a.s., Interni oddeleni, Strakonice
  - Krajska zdravotni, a.s. Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- Denmark (5):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus C
  - Bispebjerg Hospital, Copenhagen NV
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense C
- Estonia (10):
  - ECG Unit of West Tallinn Central Hospital, Tallinn, Estonia
  - West Tallinn Central Hospital, Tallinn, Estonia
  - X- Ray Department of West Tallinn Central Hospital, Tallinn, Estonia
  - X-Ray Unit, East Tallinn Central Hospital, Tallinn
  - ECG Unit, Innomedica OU and Qualitas AS (ECG Only), Tallinn
  - Innomedica OU, Tallinn
  - East Tallinn Central Hospital Internal Medical Clinic, Tallinn
  - ECG Unit, East Tallinn Central Hospital, Tallinn
  - X-Ray Department of West Tallinn Central Hospital, Tallinn
  - Mammograaf OU (Endoscopy Only), Tallinn
- France (9):
  - CHU Amiens PICARDIE - Hopital SUD, Amiens
  - Hopital Saint Andre, Bordeaux
  - Hopital Beaujon, Clichy
  - Hotel-Dieu CHU Nantes, Nantes
  - Hopital Saint Louis - Service d'hepato-gastoenterologie, Paris
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine - Service de Gastroenterologie, Paris
  - C.H.U. de Reims - Hôpital Robert Debré, Reims
  - Hopital Nord, Saint-Priest-en-Jarez
- Germany (7):
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Schlewig Holstein
  - Universitaetsmedizin Berlin, Charite Campus Virchow-Klinikum,, Berlin
  - Universitätsklinikum Halle, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Lüneburg/Abteilung Gastroenterologie, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Universitaetsklinikum Ulm, Ulm
- Hungary (12):
  - Dr Rethy Pal Korhaz-Rendelointezet, III Belgyogyaszat, Békéscsaba, Hungary
  - Szent Margit Korhaz - III Belgyogyaszat, Budapest
  - Peterfy Sandor Utcai Korhaz Rendelointezet es Baleseti Kozpont, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Belgyogyaszati Intezet Gasztroenterologiai Tanszek, Debrecen
  - Bekes Megyei Pandy Kalman Korhaz III. Gasztroenterologiai Osztaly, Gyula
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Karolina Korhaz, Mosonmagyaróvár
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, I. Sz. Belgyogyaszati Klinika, Szeged
  - Javorszky Odon Korhaz, Vác
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Beilinson campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Italy (3):
  - Istituto Clinico Humanitas IRCSS, Rozzano, Milano
  - AOR Villa Sofia-Cervello, Palermo, PA
  - AOU Mater Domini - U.O. Fisiopatologia Digestiva, Catanzaro
- Japan (20):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido P.W.F.A.C Sapporo-Kosei general Hospital, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - National Hospital Organization Mito Medical Center, Higashi-ibaraki-gun, Ibaraki
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Kuniyoshi Hospital, Kochi, Kochi
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Osaka City University Hospital, Osaka, Osaka
  - Osaka Medical College Hospital, Takatsuki-shi, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Tokyo Medical And Dental University Hospital, Faculty of Medicine, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital, Hachiōji, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Chiba University Hospital, Chiba
  - Toho University Sakura Medical Center, Chiba
  - Kurume University Hospital, Fukuoka
- Latvia (3):
  - ECG room Clinic Linezers (ECG only) Riga East University Hospital, Riga
  - X-Ray Department, Clinic Linezers (radiology only), Riga
  - Digestive Diseases Center GASTRO, Riga
- Netherlands (4):
  - VU University Medical Center (VUMC), Amsterdam
  - Academic Medical Centre, Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - Leiden University Medical Center (LUMC), Leiden
- New Zealand (9):
  - Shakespeare Specialist Group, Milford, Auckland
  - Tauranga Hospital, Tauranga, Bay of Plenty
  - Christchurch Hospital, Christchurch, Canterbury
  - Auckland City Hospital, Auckland
  - Southern District Health Board, Dunedin
  - Waikato Hospital, Hamilton
  - P3 Research Limited, Wellington
  - Pacific Radiology (X-rays only), Wellington
  - Bowen Hospital, Wellington
- Poland (10):
  - Centrum Medyczne Szpital Sw. Rodziny Sp. z o. o., Lodz, Iodzkie
  - Centrum Endoskopii Zabiegowej, Poradnia Chorob Jelitowych, Szpital Uniwersytecki nr 2 im, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Klinika Chorob Wewnetrznych i Gastroenterologii z, Warsaw, Masovian Voivodeship
  - H-T. Centrum Medyczne - ENDOTERAPIA, Tychy, Silesian Voivodeship
  - Gabinet Lekarski - Janusz Rudzinski, Bydgoszcz
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Oddzial Kliniczny Gastroenterologii Ogólnej i Onkologicznej, Uniwersytecki Szpital, Lodz
  - Endoskopia Sp. Z O.O., Sopot
  - Nzoz Vivamed, Warsaw
  - Lexmedica, Wroclaw
- Romania (2):
  - Cabinet Particular Policlinic Algomed Srl, Timișoara, Timiș County
  - Spitalul Universitar de Urgenta Bucharest, Bucharest
- Russia (11):
  - Municipal Institution of Healthcare City Clinical Hospital 12,, Saratov, Russia
  - Federal state budget institution "State scientific centre of coloproctology", Moscow
  - State Budget Institution of Healthcare Nizhniy Novgorod Regional Clinical Hospital named after N. A., Nizhny Novgorod
  - Federal state Institution "Sibirian regional Medical centre of Federal Medicobiologic Agency",, Novosibirsk
  - Municipal Budget Institution of Healthcare of Novosibirsk " City Clinical Hospital No 12", Novosibirsk
  - State Budget Educational Institution of Higher Professional Education, Novosibirsk
  - Federal State Budgetary Institution "Scientific Research Institute of Physiology and Fundamental, Novosibirsk
  - Non-State Healthcare Institution "Road Clinical Hospital at the station Samara", Samara
  - Limited Liability Company Medical Company "Hepatolog", Samara
  - Samara Diagnostic center, X-ray Department, Samara
  - State budget institution of healthcare of Yaroslavl region Regional clinical hospital, Yaroslavl
- Serbia (7):
  - Clinical Centre of Serbia, Clinic for Gastroenterology and Hepatology, Belgrade, Serbia, Europe
  - Clinical Hospital Centre Zvezdara, Belgrade
  - Military Medical Academy Belgrade, Belgrade
  - Clinical Centre of Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Clinic for Gastroenterology and Hepatology, Novi Sad
  - Clinical Centre of Vojvodina, Emergency Internal Medicine Division, Novi Sad
  - "General Hospital ""Djordje Joanovic"", Zrenjanin
- Slovakia (4):
  - Medak s.r.o., Bratislava
  - KM Management spol. s.r.o., Nitra
  - Aura SA, s.r.o., Nové Mesto nad Váhom
  - Gastro I., s.r.o., Prešov
- South Africa (5):
  - Dr John Philip Wright, Claremont, Cape Town
  - Chris Hani Baragwanath Academic Hospital, Johannesburg, Gauteng
  - Panorama MediClinic, Cape Town, Western Cape
  - Louis Leipoldt Medical Centre, Cape Town, Western Cape
  - Endocare Research Centre, Western Cape
- South Korea (6):
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - KyungHee University Hospital, Seoul, Republic of Korea
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital,, Seoul
- Spain (4):
  - Hospital Universitari de Bellvitge, Servicio de Digestivo, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
- National Taiwan University Hospital, Taipei, Taiwan
- Ukraine (16):
  - Internal Medicine Center of Crimean Republic Institution"Clinical Territorial Medical Community", Simferopol, Ar Krym
  - Municipal Healthcare Institution Kharkiv City Clinical Hospital #2, Proctology Department, Kharkiv, Ukraine
  - SI "Railway Hospital of the SI "Odesa Railway"", Polyclinic Department,, Odesa, Ukraine
  - Regional Municipal Institution "Chernivtsi Regional Clinical Hospital", Chernivtsi
  - Regional Municipal Institution Chernivtsi Regional Clinical Hospital,, Chernivtsi
  - State Institution "Institute of Gastroenterology of the National Academy of Medical Sciences of, Dniepropetrovsk
  - State Institution "National L.T. Malaya Therapy Institute of National Academy of, Kharkiv
  - Kyiv Municipal Clinical Hospital #18, Proctology Department, Kyiv
  - LTD "St. Paraskeva Medical Center", Lviv
  - Municipal City Clinical Hospital of the Emergency Medical Care, 1-st Therapy Department of hospital,, Lviv
  - Municipal Institution "Odesa Regional Clinical Hospital", Odesa
  - SI "District Clin. Hosp.of Uzhgorod station (STSA "Lviv Railway", Therapy Dep., SBHEI "Uzhgorod Nat., Uzhhorod
  - Vinnytsia Regional Clinical Hospital for Invalids of the Great Patriotic War, Therapy Department #2,, Vinnytsia
  - Motor-Sich clinic, LLC, Zaporizhzhia
  - Minicipal Institution City Hospital 7, Therapevtic Department,, Zaporizhzhia
  - Municipal Institution "City Hospital #7", Zaporizhzhia State Medical University, Zaporizhzhia
- United Kingdom (7):
  - Addenbrooke's Hospital-Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Department of Gastroenterology, Old Building, Bristol, England
  - University College Hospital, London, Greater London
  - NWLH NHS trust, Harrow, Middlesex
  - The North West London Hospitals NHS Trust, Harrow, Middlesex
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Addenbrooke's Hospital, Cambridge

REFERENCES:
- [Derived] Panes J, D'Haens GR, Sands BE, Ng SC, Lawendy N, Kulisek N, Guo X, Wu J, Vranic I, Panaccione R, Vermeire S. Analysis of tofacitinib safety in ulcerative colitis from the completed global clinical developmental program up to 9.2 years of drug exposure. United European Gastroenterol J. 2024 Jul;12(6):793-801. doi: 10.1002/ueg2.12584. Epub 2024 May 22. PMID 38778549
- [Derived] Rubin DT, Torres J, Regueiro M, Reinisch W, Prideaux L, Kotze PG, Tan FH, Gardiner S, Mundayat R, Cadatal MJ, Ng SC. Association Between Smoking Status and the Efficacy and Safety of Tofacitinib in Patients with Ulcerative Colitis. Crohns Colitis 360. 2024 Jan 20;6(1):otae004. doi: 10.1093/crocol/otae004. eCollection 2024 Jan. PMID 38425446
- [Derived] Rubin DT, Salese L, Cohen M, Kotze PG, Woolcott JC, Su C, Mundayat R, Paulissen J, Torres J, Long MD. Presence of risk factors associated with colectomy among patients with ulcerative colitis: a post hoc analysis of data from the tofacitinib OCTAVE ulcerative colitis clinical program. Therap Adv Gastroenterol. 2023 Aug 7;16:17562848231189122. doi: 10.1177/17562848231189122. eCollection 2023. PMID 37560161
- [Derived] Schreiber S, Rubin DT, Ng SC, Peyrin-Biroulet L, Danese S, Modesto I, Guo X, Su C, Kwok KK, Jo H, Chen Y, Yndestad A, Reinisch W, Dubinsky MC. Major Adverse Cardiovascular Events by Baseline Cardiovascular Risk in Patients with Ulcerative Colitis Treated with Tofacitinib: Data from the OCTAVE Clinical Programme. J Crohns Colitis. 2023 Nov 24;17(11):1761-1770. doi: 10.1093/ecco-jcc/jjad104. PMID 37402275
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Lee SD, Allegretti JR, Steinwurz F, Connelly SB, Lawendy N, Paulissen J, Gecse KB. Tofacitinib as a maintenance therapy in patients with ulcerative colitis stratified by OCTAVE Sustain baseline Mayo endoscopic subscore. BMC Gastroenterol. 2023 Feb 8;23(1):34. doi: 10.1186/s12876-022-02508-2. PMID 36755231
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Sandborn WJ, Sands BE, Vermeire S, Leung Y, Guo X, Modesto I, Su C, Wang W, Panes J. Modified Mayo score versus Mayo score for evaluation of treatment efficacy in patients with ulcerative colitis: data from the tofacitinib OCTAVE program. Therap Adv Gastroenterol. 2022 Dec 5;15:17562848221136331. doi: 10.1177/17562848221136331. eCollection 2022. PMID 36506749
- [Derived] Lichtenstein GR, Bressler B, Francisconi C, Vermeire S, Lawendy N, Salese L, Sawyerr G, Shi H, Su C, Judd DT, Jones T, Loftus EV. Assessment of Safety and Efficacy of Tofacitinib, Stratified by Age, in Patients from the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):27-41. doi: 10.1093/ibd/izac084. PMID 36342120
- [Derived] Hudesman DP, Torres J, Salese L, Woolcott JC, Mundayat R, Su C, Mosli MH, Allegretti JR. Long-Term Improvement in the Patient-Reported Outcomes of Rectal Bleeding, Stool Frequency, and Health-Related Quality of Life with Tofacitinib in the Ulcerative Colitis OCTAVE Clinical Program. Patient. 2023 Mar;16(2):95-103. doi: 10.1007/s40271-022-00603-w. Epub 2022 Nov 7. PMID 36336750
- [Derived] Targownik L, Dubinsky MC, Steinwurz F, Bushmakin AG, Cappelleri JC, Tai E, Gardiner S, Hur P, Panes J. Disease Activity and Health-related Quality of Life Relationships with Work Productivity in Patients with Ulcerative Colitis in OCTAVE Induction 1 and 2 and OCTAVE Sustain. J Crohns Colitis. 2023 Apr 19;17(4):513-523. doi: 10.1093/ecco-jcc/jjac161. PMID 36271912
- [Derived] Sandborn WJ, D'Haens GR, Sands BE, Panaccione R, Ng SC, Lawendy N, Kulisek N, Modesto I, Guo X, Mundayat R, Su C, Vranic I, Panes J. Tofacitinib for the Treatment of Ulcerative Colitis: An Integrated Summary of up to 7.8 Years of Safety Data from the Global Clinical Programme. J Crohns Colitis. 2023 Apr 3;17(3):338-351. doi: 10.1093/ecco-jcc/jjac141. PMID 36124702
- [Derived] Loftus EV, Baumgart DC, Gecse K, Kinnucan JA, Connelly SB, Salese L, Su C, Kwok KK, Woolcott JC, Armuzzi A. Clostridium difficile Infection in Patients with Ulcerative Colitis Treated with Tofacitinib in the Ulcerative Colitis Program. Inflamm Bowel Dis. 2023 May 2;29(5):744-751. doi: 10.1093/ibd/izac139. PMID 35792493
- [Derived] Winthrop KL, Vermeire S, Long MD, Panes J, Ng SC, Kulisek N, Mundayat R, Lawendy N, Vranic I, Modesto I, Su C, Melmed GY. Long-term Risk of Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2023 Jan 5;29(1):85-96. doi: 10.1093/ibd/izac063. PMID 35648151
- [Derived] Vavricka SR, Greuter T, Cohen BL, Reinisch W, Steinwurz F, Fellmann M, Guo X, Lawendy N, Paulissen J, Peyrin-Biroulet L. Corticosteroid-free efficacy and safety outcomes in patients receiving tofacitinib in the OCTAVE Sustain maintenance study. Therap Adv Gastroenterol. 2022 May 10;15:17562848221090834. doi: 10.1177/17562848221090834. eCollection 2022. PMID 35574426
- [Derived] Mukherjee A, Tsuchiwata S, Nicholas T, Cook JA, Modesto I, Su C, D'Haens GR, Sandborn WJ. Exposure-Response Characterization of Tofacitinib Efficacy in Moderate to Severe Ulcerative Colitis: Results From Phase II and Phase III Induction and Maintenance Studies. Clin Pharmacol Ther. 2022 Jul;112(1):90-100. doi: 10.1002/cpt.2601. Epub 2022 Apr 27. PMID 35380740
- [Derived] Feagan BG, Khanna R, Sandborn WJ, Vermeire S, Reinisch W, Su C, Salese L, Fan H, Paulissen J, Woodworth DA, Niezychowski W, Sands BE. Agreement between local and central reading of endoscopic disease activity in ulcerative colitis: results from the tofacitinib OCTAVE trials. Aliment Pharmacol Ther. 2021 Dec;54(11-12):1442-1453. doi: 10.1111/apt.16626. Epub 2021 Oct 6. PMID 34614208
- [Derived] Farraye FA, Qazi T, Kotze PG, Moore GT, Mundayat R, Lawendy N, Sharma PP, Judd DT. The impact of body mass index on efficacy and safety in the tofacitinib OCTAVE ulcerative colitis clinical programme. Aliment Pharmacol Ther. 2021 Aug;54(4):429-440. doi: 10.1111/apt.16439. Epub 2021 Jun 24. PMID 34165201
- [Derived] Rubin DT, Reinisch W, Greuter T, Kotze PG, Pinheiro M, Mundayat R, Maller E, Fellmann M, Lawendy N, Modesto I, Vavricka SR, Lichtenstein GR. Extraintestinal manifestations at baseline, and the effect of tofacitinib, in patients with moderate to severe ulcerative colitis. Therap Adv Gastroenterol. 2021 May 16;14:17562848211005708. doi: 10.1177/17562848211005708. eCollection 2021. PMID 34035832
- [Derived] Panes J, Vermeire S, Dubinsky MC, Loftus EV, Lawendy N, Wang W, Salese L, Su C, Modesto I, Guo X, Colombel JF. Efficacy and Safety of Tofacitinib Re-treatment for Ulcerative Colitis After Treatment Interruption: Results from the OCTAVE Clinical Trials. J Crohns Colitis. 2021 Nov 8;15(11):1852-1863. doi: 10.1093/ecco-jcc/jjab065. PMID 33884415
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Sharara AI, Su C, Modesto I, Mundayat R, Gunay LM, Salese L, Sands BE. Efficacy and Safety of Tofacitinib in Ulcerative Colitis Based on Prior Tumor Necrosis Factor Inhibitor Failure Status. Clin Gastroenterol Hepatol. 2022 Mar;20(3):591-601.e8. doi: 10.1016/j.cgh.2021.02.043. Epub 2021 Mar 6. PMID 33684552
- [Derived] Vong C, Martin SW, Deng C, Xie R, Ito K, Su C, Sandborn WJ, Mukherjee A. Population Pharmacokinetics of Tofacitinib in Patients With Moderate to Severe Ulcerative Colitis. Clin Pharmacol Drug Dev. 2021 Mar;10(3):229-240. doi: 10.1002/cpdd.899. Epub 2021 Jan 29. PMID 33513294
- [Derived] Curtis JR, Regueiro M, Yun H, Su C, DiBonaventura M, Lawendy N, Nduaka CI, Koram N, Cappelleri JC, Chan G, Modesto I, Lichtenstein GR. Tofacitinib Treatment Safety in Moderate to Severe Ulcerative Colitis: Comparison of Observational Population Cohort Data From the IBM MarketScan(R) Administrative Claims Database With Tofacitinib Trial Data. Inflamm Bowel Dis. 2021 Aug 19;27(9):1394-1408. doi: 10.1093/ibd/izaa289. PMID 33324993
- [Derived] Colombel JF, Osterman MT, Thorpe AJ, Salese L, Nduaka CI, Zhang H, Lawendy N, Friedman GS, Quirk D, Su C, Reinisch W. Maintenance of Remission With Tofacitinib Therapy in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2022 Jan;20(1):116-125.e5. doi: 10.1016/j.cgh.2020.10.004. Epub 2020 Oct 9. PMID 33039585
- [Derived] Sands BE, Colombel JF, Ha C, Farnier M, Armuzzi A, Quirk D, Friedman GS, Kwok K, Salese L, Su C, Taub PR. Lipid Profiles in Patients With Ulcerative Colitis Receiving Tofacitinib-Implications for Cardiovascular Risk and Patient Management. Inflamm Bowel Dis. 2021 May 17;27(6):797-808. doi: 10.1093/ibd/izaa227. PMID 32870265
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Lichtenstein GR, Rogler G, Ciorba MA, Su C, Chan G, Pedersen RD, Lawendy N, Quirk D, Nduaka CI, Thorpe AJ, Panes J. Tofacitinib, an Oral Janus Kinase Inhibitor: Analysis of Malignancy (Excluding Nonmelanoma Skin Cancer) Events Across the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2021 May 17;27(6):816-825. doi: 10.1093/ibd/izaa199. PMID 32766762
- [Derived] Sandborn WJ, Panes J, Sands BE, Reinisch W, Su C, Lawendy N, Koram N, Fan H, Jones TV, Modesto I, Quirk D, Danese S. Venous thromboembolic events in the tofacitinib ulcerative colitis clinical development programme. Aliment Pharmacol Ther. 2019 Nov;50(10):1068-1076. doi: 10.1111/apt.15514. Epub 2019 Oct 9. PMID 31599001
- [Derived] Sands BE, Taub PR, Armuzzi A, Friedman GS, Moscariello M, Lawendy N, Pedersen RD, Chan G, Nduaka CI, Quirk D, Salese L, Su C, Feagan BG. Tofacitinib Treatment Is Associated With Modest and Reversible Increases in Serum Lipids in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2020 Jan;18(1):123-132.e3. doi: 10.1016/j.cgh.2019.04.059. Epub 2019 May 8. PMID 31077827
- [Derived] Sandborn WJ, Panes J, D'Haens GR, Sands BE, Su C, Moscariello M, Jones T, Pedersen R, Friedman GS, Lawendy N, Chan G. Safety of Tofacitinib for Treatment of Ulcerative Colitis, Based on 4.4 Years of Data From Global Clinical Trials. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1541-1550. doi: 10.1016/j.cgh.2018.11.035. Epub 2018 Nov 23. PMID 30476584
- [Derived] Winthrop KL, Melmed GY, Vermeire S, Long MD, Chan G, Pedersen RD, Lawendy N, Thorpe AJ, Nduaka CI, Su C. Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2018 Sep 15;24(10):2258-2265. doi: 10.1093/ibd/izy131. PMID 29850873
- [Derived] Motoya S, Watanabe M, Kim HJ, Kim YH, Han DS, Yuasa H, Tabira J, Isogawa N, Arai S, Kawaguchi I, Hibi T. Tofacitinib induction and maintenance therapy in East Asian patients with active ulcerative colitis: subgroup analyses from three phase 3 multinational studies. Intest Res. 2018 Apr;16(2):233-245. doi: 10.5217/ir.2018.16.2.233. Epub 2018 Apr 30. PMID 29743836
- [Derived] Panes J, Vermeire S, Lindsay JO, Sands BE, Su C, Friedman G, Zhang H, Yarlas A, Bayliss M, Maher S, Cappelleri JC, Bushmakin AG, Rubin DT. Tofacitinib in Patients with Ulcerative Colitis: Health-Related Quality of Life in Phase 3 Randomised Controlled Induction and Maintenance Studies. J Crohns Colitis. 2018 Jan 24;12(2):145-156. doi: 10.1093/ecco-jcc/jjx133. PMID 29028981
- [Derived] Sandborn WJ, Su C, Sands BE, D'Haens GR, Vermeire S, Schreiber S, Danese S, Feagan BG, Reinisch W, Niezychowski W, Friedman G, Lawendy N, Yu D, Woodworth D, Mukherjee A, Zhang H, Healey P, Panes J; OCTAVE Induction 1, OCTAVE Induction 2, and OCTAVE Sustain Investigators. Tofacitinib as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2017 May 4;376(18):1723-1736. doi: 10.1056/NEJMoa1606910. PMID 28467869
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921096&StudyName=A%20Study%20Of%20Oral%20CP-690%2C550%20As%20A%20Maintenance%20Therapy%20For%20Ulcerative%20Colitis

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib 5 mg BID: Participants received tofacitinib (CP-690,550) 5 mg tablets, orally, BID for 53 weeks of double blind treatment period. Participants were followed-up for 4 weeks if withdrew from study participation.
- Tofacitinib 10 mg BID: Participants received tofacitinib 10 mg tablets, orally, BID for 53 weeks of double blind treatment period. Participants were followed-up for 4 weeks if withdrew from study participation.
- Placebo: Participants received tofacitinib matched placebo tablets, orally, BID for 53 weeks of double blind treatment period. Participants were followed-up for 4 weeks if withdrew from study participation.
Period: Overall Study
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Started | 198 | 197 | 198
Treated | 198 | 196 | 198
Completed | 111 | 126 | 53
Not Completed | 87 | 71 | 145
Not completed — Adverse Event | 5 | 9 | 7
Not completed — Lack of Efficacy | 70 | 53 | 132
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — Pregnancy | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 5
Not completed — Other | 2 | 1 | 0
Not completed — Randomized but not treated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo | Total
Number analyzed (Participants) | 198 | 197 | 198 | 593
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (13.7) | 42.9 (14.4) | 43.4 (14) | 42.7 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 87 | 82 | 264
  Male | 103 | 110 | 116 | 329

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants In Remission at Week 52
Description: Remission in participants was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of ulcerative colitis (UC). It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and physician global assessment (PGA), each subscore graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12 where higher score indicating higher disease severity.
Time Frame: Week 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 34.3 | 40.6 | 11.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; P-value based on Cochran-Mantel-Haenszel (CMH) chi-square test stratified by induction study treatment and baseline remission status. Difference and its 95 percent (%) confidence interval (CI) based on normal approximation for the difference in binomial proportions. Missing data were imputed using Non-responder imputation (NRI); Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 23.2, 95% CI 2-sided [15.3 to 31.2]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; P-value based on CMH chi-square test stratified by induction study treatment and baseline remission status. Difference and its 95% CI based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 29.5, 95% CI 2-sided [21.4 to 37.6]

2. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 52
Description: Mucosal healing in participants was defined by mayo endoscopic subscore of 0 or 1. The mayo endoscopic subscore consisted of the findings of centrally read flexible sigmoidoscopy, graded from 0 to 3 with higher subscores indicating higher disease severity.
Time Frame: Week 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 37.4 | 45.7 | 13.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 24.2, 95% CI 2-sided [16.0 to 32.5]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 32.6, 95% CI 2-sided [24.2 to 41.0]

3. Secondary Outcome: Percentage of Participants With Sustained Steroid-Free Remission (Defined as Being in Remission and Steroid-Free at Both Week 24 and 52), Among Participants With Remission at Baseline
Description: Sustained steroid-free remission was defined by being in remission and steroid-free at both Week 24 and Week 52. Steroid-free remission was defined by being in remission, in addition to no requirement of any treatment with steroid for at least 4 weeks prior to the visit. Remission was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity. Percentage of participants with sustained steroid-free remission (among participants with remission at baseline) were reported in this outcome measure.
Time Frame: Week 24, 52
Population: FAS included all randomized participants. Here "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 65 | 55 | 59
percentage of participants | 35.4 | 47.3 | 5.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; P-value based on CMH chi-square test stratified by induction study treatment. Difference and its 95% CI based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 30.3, 95% CI 2-sided [17.4 to 43.2]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 42.2, 95% CI 2-sided [27.9 to 56.5]

4. Secondary Outcome: Percentage of Participants in Remission at Week 24
Description: Remission in participants was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher subscores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity.
Time Frame: Week 24
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 33.8 | 35.5 | 11.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 22.7, 95% CI 2-sided [14.8 to 30.6]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 24.4, 95% CI 2-sided [16.4 to 32.4]

5. Secondary Outcome: Percentage of Participants in Sustained Remission
Description: Sustained remission in participants was defined by being in remission at both Week 24 and Week 52. Remission was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher subscores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher score indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 22.2 | 25.4 | 5.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 17.2, 95% CI 2-sided [10.6 to 23.7]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 20.3, 95% CI 2-sided [13.5 to 27.1]

6. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 24
Description: Mucosal healing in participants was defined by a mayo endoscopic subscore of 0 or 1. The mayo endoscopic subscore consisted of the findings of centrally read flexible sigmoidoscopy, graded from 0 to 3 with higher scores indicating higher disease severity.
Time Frame: Week 24
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 43.9 | 46.2 | 17.2
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 26.8, 95% CI 2-sided [18.1 to 35.5]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 29.0, 95% CI 2-sided [20.3 to 37.7]

7. Secondary Outcome: Percentage of Participants With Sustained Mucosal Healing
Description: Sustained mucosal healing in participants was defined by achieving mayo endoscopic subscore of 0 or 1 at both Week 24 and Week 52. The mayo endoscopic subscore consisted of the findings of centrally read flexible sigmoidoscopy, graded from 0 to 3 with higher scores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 27.8 | 33.0 | 6.6
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 21.2, 95% CI 2-sided [14.1 to 28.3]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 26.4, 95% CI 2-sided [19.0 to 33.8]

8. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 24 and 52, Among Participants With Mucosal Healing at Baseline
Description: Mucosal healing in participants was defined as achieving mayo endoscopic subscore of 0 or 1. The mayo endoscopic subscore consisted of the findings of centrally read flexible sigmoidoscopy, graded from 0 to 3 with higher scores indicating higher disease severity.
Time Frame: Week 24, 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 105 | 89 | 101
percentage of participants
  Week 24 | 52.4 | 66.3 | 21.8
  Week 52 | 41.9 | 55.1 | 11.9
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; At Week 24: P-value based on CMH chi-square test stratified by induction study treatment. Difference and its 95% CI based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 30.6, 95% CI 2-sided [18.1 to 43.1]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 44.5, 95% CI 2-sided [31.8 to 57.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; At Week 52: P-value based on CMH chi-square test stratified by induction study treatment. Difference and its 95% CI based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 30.0, 95% CI 2-sided [18.7 to 41.4]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 43.2, 95% CI 2-sided [31.1 to 55.3]

9. Secondary Outcome: Percentage of Participants With Sustained Mucosal Healing, Among Participants With Mucosal Healing at Baseline
Description: as for outcome 7
Time Frame: Week 24, 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 105 | 89 | 101
percentage of participants | 33.3 | 49.4 | 8.9
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 24.4, 95% CI 2-sided [13.8 to 35.0]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 40.5, 95% CI 2-sided [28.7 to 52.3]

10. Secondary Outcome: Percentage of Participants With Clinical Response at Week 24 and 52
Description: Clinical response was defined by a decrease from induction study (A3921094 [NCT01465763] or A3921095 [NCT01458951]) baseline in Mayo score of at least 3 points and at least 30%, with an accompanying decrease in the rectal bleeding subscore of at least 1 point, or an absolute rectal bleeding subscore of 0 or 1. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity. Percentage of participants with clinical response at Week 24 and 52 have been reported in this outcome measure.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants
  Week 24 | 63.6 | 70.6 | 33.3
  Week 52 | 51.5 | 61.9 | 20.2
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; At Week 24: P-value based on CMH chi-square test stratified by induction study treatment and baseline remission status. Difference and its 95% CI based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 30.3, 95% CI 2-sided [20.9 to 39.7]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 37.2, 95% CI 2-sided [28.1 to 46.4]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; At Week 52: P-value based on CMH chi-square test stratified by induction study treatment and baseline remission status. Difference and its 95% CI based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 31.3, 95% CI 2-sided [22.4 to 40.2]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 41.7, 95% CI 2-sided [32.9 to 50.5]

11. Secondary Outcome: Percentage of Participants With Sustained Clinical Response
Description: Sustained clinical response in participants was defined as showing clinical response at both Week 24 and Week 52. Clinical response was defined by a decrease from induction study (A3921094 [NCT01465763] or A3921095 [NCT01458951]) baseline in mayo score of at least 3 points and at least 30%, with an accompanying decrease in the rectal bleeding subscore of at least 1 point, or an absolute rectal bleeding subscore of 0 or 1. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity. Percentage of participants with sustained clinical response are reported in this outcome measure.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 49.0 | 59.4 | 19.2
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 29.8, 95% CI 2-sided [20.9 to 38.7]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 40.2, 95% CI 2-sided [31.4 to 49.0]

12. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 24 and 52
Description: Clinical remission in participants was defined as a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants
  Week 24 | 34.3 | 35.5 | 11.1
  Week 52 | 34.3 | 41.1 | 11.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 23.2, 95% CI 2-sided [15.3 to 31.2]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 24.4, 95% CI 2-sided [16.4 to 32.4]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 23.2, 95% CI 2-sided [15.3 to 31.2]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 30.0, 95% CI 2-sided [21.9 to 38.2]

13. Secondary Outcome: Percentage of Participants in Sustained Clinical Remission
Description: Sustained clinical remission in participants was defined as being in clinical remission at both Week 24 and Week 52. Clinical remission was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 22.2 | 25.9 | 5.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 17.2, 95% CI 2-sided [10.6 to 23.7]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 20.8, 95% CI 2-sided [14.0 to 27.7]

14. Secondary Outcome: Percentage of Participants in Deep Remission at Week 24 and 52
Description: Deep remission in participants was defined as a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and 0 subscore for both rectal bleeding and endoscopic subscores. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants
  Week 24 | 14.1 | 10.7 | 4.0
  Week 52 | 14.6 | 15.2 | 4.0
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.0006, CMH chi-square test; Difference in percentage = 10.1, 95% CI 2-sided [4.5 to 15.7]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.0092, CMH chi-square test; Difference in percentage = 6.6, 95% CI 2-sided [1.5 to 11.7]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.0004, CMH chi-square test; Difference in percentage = 10.6, 95% CI 2-sided [5.0 to 16.2]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 11.2, 95% CI 2-sided [5.5 to 16.9]

15. Secondary Outcome: Percentage of Participants in Sustained Deep Remission
Description: Sustained deep remission was defined by being in deep remission at both Week 24 and Week 52. Deep remission in participants was defined as a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and 0 subscore for both rectal bleeding and endoscopic subscores. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 6.1 | 3.6 | 0.5
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0029, CMH chi-square test; Difference in percentage = 5.6, 95% CI 2-sided [2.1 to 9.0]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0350, CMH chi-square test; Difference in percentage = 3.0, 95% CI 2-sided [0.3 to 5.8]

16. Secondary Outcome: Percentage of Participants in Symptomatic Remission at Week 24 and 52
Description: Symptomatic remission in participants was defined as a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point, and 0 subscore for both rectal bleeding and stool frequency. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 sub-scores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants
  Week 24 | 23.7 | 21.8 | 6.6
  Week 52 | 22.7 | 26.9 | 7.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 17.2, 95% CI 2-sided [10.3 to 24.0]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 15.3, 95% CI 2-sided [8.5 to 22.0]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 15.7, 95% CI 2-sided [8.8 to 22.5]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 19.8, 95% CI 2-sided [12.7 to 27.0]

17. Secondary Outcome: Percentage of Participants in Sustained Symptomatic Remission
Description: Sustained symptomatic remission in participants was defined as being in symptomatic remission at both Week 24 and Week 52. Symptomatic remission was defined as a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point, and 0 subscore for both rectal bleeding and stool frequency. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 13.6 | 15.7 | 2.5
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 11.1, 95% CI 2-sided [5.9 to 16.4]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 13.2, 95% CI 2-sided [7.7 to 18.7]

18. Secondary Outcome: Percentage of Participants in Endoscopic Remission at Week 24 and 52
Description: Endoscopic remission in participants was defined as a mayo endoscopic subscore of 0. The mayo endoscopic subscore consisted of the findings of centrally read flexible sigmoidoscopy, graded from 0 to 3 with higher subscores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants
  Week 24 | 16.2 | 12.2 | 4.0
  Week 52 | 14.6 | 16.8 | 4.0
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 12.1, 95% CI 2-sided [6.3 to 17.9]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.0021, CMH chi-square test; Difference in percentage = 8.1, 95% CI 2-sided [2.8 to 13.5]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.0004, CMH chi-square test; Difference in percentage = 10.6, 95% CI 2-sided [5.0 to 16.2]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 12.7, 95% CI 2-sided [6.8 to 18.6]

19. Secondary Outcome: Percentage of Participants in Sustained Endoscopic Remission
Description: Sustained endoscopic remission in participants was defined as being in endoscopic remission at both Week 24 and Week 52. Endoscopic remission was defined by a mayo endoscopic subscore of 0. The mayo endoscopic subscore consisted of the findings of centrally read flexible sigmoidoscopy, graded from 0 to 3 with higher subscores indicating higher disease severity.
Time Frame: Week 24, 52
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
percentage of participants | 6.1 | 5.1 | 0.5
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0029, CMH chi-square test; Difference in percentage = 5.6, 95% CI 2-sided [2.1 to 9.0]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0064, CMH chi-square test; Difference in percentage = 4.6, 95% CI 2-sided [1.4 to 7.8]

20. Secondary Outcome: Total Mayo Score at Baseline, Week 24 and 52
Description: Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity.
Time Frame: Baseline, Week 24, 52
Population: FAS included all randomized participants. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
units on a scale
  Baseline (n = 198, 197, 198) | 3.3 (1.8) | 3.4 (1.8) | 3.3 (1.8)
  Week 24 (n = 179, 186, 181) | 4.1 (3.4) | 4.0 (3.3) | 6.7 (3.5)
  Week 52 (n = 129, 137, 68) | 3.2 (3.1) | 2.6 (2.7) | 4.6 (3.2)

21. Secondary Outcome: Change From Baseline in Total Mayo Score at Week 24 and 52
Description: Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity. Change from baseline in total mayo score at Week 24 and 52 was reported.
Time Frame: Baseline, Week 24, 52
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 198 | 197 | 198
units on a scale
  Change at Week 24 (n = 179, 186, 181) | 0.3 (0.3) | 0.0 (0.3) | 2.9 (0.3)
  Change at Week 52 (n = 129, 137, 68) | 0.4 (0.3) | -0.4 (0.3) | 2.9 (0.4)
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; At Week 24; Test type: Superiority or Other; p < 0.0001, Linear mixed effect model; Least Square Mean Difference = -2.6, 95% CI 2-sided [-3.2 to -1.9]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; At Week 24; Test type: Superiority or Other; p < 0.0001, Linear mixed effect model; Least Square Mean Difference = -2.8, 95% CI 2-sided [-3.5 to -2.2]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; At Week 52; Test type: Superiority or Other; p < 0.0001, Linear mixed effect model; Least Square Mean Difference = -2.6, 95% CI 2-sided [-3.4 to -1.7]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; At Week 52; Test type: Superiority or Other; p < 0.0001, Linear mixed effect model; Least Square Mean Difference = -3.3, 95% CI 2-sided [-4.1 to -2.5]

22. Secondary Outcome: Percentage of Participants in Remission, Among Participants With Remission at Baseline
Description: Remission in participants was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher score indicating higher disease severity.
Time Frame: Week 24, 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 65 | 55 | 59
percentage of participants
  Week 24 | 55.4 | 63.6 | 15.3
  Week 52 | 46.2 | 56.4 | 10.2
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 40.1, 95% CI 2-sided [25.0 to 55.3]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 48.4, 95% CI 2-sided [32.7 to 64.1]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 36.0, 95% CI 2-sided [21.6 to 50.3]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 46.2, 95% CI 2-sided [31.0 to 61.4]

23. Secondary Outcome: Percentage of Participants in Sustained Remission, Among Participants With Remission at Baseline
Description: Sustained remission in participants was defined by being in remission at both Week 24 and Week 52. Remission was defined as a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher score indicating higher disease severity.
Time Frame: Week 24, 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 65 | 55 | 59
percentage of participants | 36.9 | 47.3 | 5.1
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 31.8, 95% CI 2-sided [18.8 to 44.8]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 42.2, 95% CI 2-sided [27.9 to 56.5]

24. Secondary Outcome: Percentage of Participants in Steroid-free Remission, Among Participants in Remission at Baseline
Description: Steroid-free remission was defined by being in remission, in addition to no requirement of any treatment with steroid for at least 4 weeks prior to the visit. Remission was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity. Percentage of participants in steroid-free remission were reported in this outcome measure.
Time Frame: Week 24, 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 65 | 55 | 59
percentage of participants
  Week 24 | 53.8 | 63.6 | 15.3
  Week 52 | 44.6 | 56.4 | 10.2
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 38.6, 95% CI 2-sided [23.4 to 53.8]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 48.4, 95% CI 2-sided [32.7 to 64.1]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 34.4, 95% CI 2-sided [20.1 to 48.8]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.0001, CMH chi-square test; Difference in percentage = 46.2, 95% CI 2-sided [31.0 to 61.4]

25. Secondary Outcome: Percentage of Participants in Steroid-Free Remission, Among Participants Receiving Steroids at Baseline
Description: Steroid-free remission was defined by being in remission, in addition to no requirement of any treatment with steroid for at least 4 weeks prior to the visit. Remission was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity. Percentage of participants with steroid-free remission were reported in this outcome measure.
Time Frame: Week 24, 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 101 | 87 | 101
percentage of participants
  Week 24 | 23.8 | 24.1 | 10.9
  Week 52 | 27.7 | 27.6 | 10.9
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.0074, CMH chi-square test; Difference in percentage = 12.9, 95% CI 2-sided [2.6 to 23.2]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.0103, CMH chi-square test; Difference in percentage = 13.2, 95% CI 2-sided [2.4 to 24.1]
Statistical Analysis 3: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.0018, CMH chi-square test; Difference in percentage = 16.8, 95% CI 2-sided [6.2 to 27.5]
Statistical Analysis 4: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.0029, CMH chi-square test; Difference in percentage = 16.7, 95% CI 2-sided [5.5 to 27.9]

26. Secondary Outcome: Percentage of Participants in Sustained Steroid-Free Remission, Among Participants Receiving Steroids at Baseline
Description: Sustained steroid-free remission was defined by being in remission and steroid-free at both Week 24 and Week 52. Steroid-free remission was defined by being in remission, in addition to no requirement of any treatment with steroid for at least 4 weeks prior to the visit. Remission was defined by a total mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating higher disease severity. These subscores were summed up to give a total score range of 0 to 12, where higher scores indicating higher disease severity. Percentage of participants with sustained steroid-free remission were reported in this outcome measure.
Time Frame: Week 24, 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Number analyzed (Participants) | 101 | 87 | 101
percentage of participants | 12.9 | 16.1 | 5.0
Statistical Analysis 1: Comparison: Tofacitinib 5 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0419, CMH chi-square test; Difference in percentage = 7.9, 95% CI 2-sided [0.1 to 15.7]
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0121, CMH chi-square test; Difference in percentage = 11.1, 95% CI 2-sided [2.3 to 19.9]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 57
Description: Same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis included all treated participants.
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 10/198 | 11/196 | 13/198
Other Adverse Events (participants affected / at risk) | 87/198 | 107/196 | 108/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tofacitinib 5 mg BID (N=198) | Tofacitinib 10 mg BID (N=196) | Placebo (N=198)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/95 | 0/86 | 1/82 — This AE was gender specific.
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/95 | 0/86 | 0/82 — This AE was gender specific.
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=198) | Tofacitinib 10 mg BID (N=196) | Placebo (N=198)
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 11
Colitis ulcerative (Gastrointestinal disorders) | 35 | 29 | 64
Fatigue (General disorders) | 8 | 4 | 11
Herpes zoster (Infections and infestations) | 2 | 10 | 1
Nasopharyngitis (Infections and infestations) | 19 | 27 | 11
Upper respiratory tract infection (Infections and infestations) | 13 | 12 | 7
Blood creatine phosphokinase increased (Investigations) | 6 | 13 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 11 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 17 | 19
Headache (Nervous system disorders) | 17 | 6 | 12
Rash (Skin and subcutaneous tissue disorders) | 6 | 11 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.